CLINICAL TRIAL: NCT00091988
Title: Program to Reduce Incontinence by Diet and Exercise
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01DK067860 (NIH); U01DK067860 (NIH)
Record Dates: First submitted 2004-09-21; First posted 2004-09-22 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Weight Loss; Obesity; Motivation
MeSH Terms: conditions — Urinary Incontinence; Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle & Behavioral Change Program (Experimental)
  Interventions: Behavioral: Lifestyle & Behavioral Change Program
- Structured Education Program (Active Comparator)
  Interventions: Behavioral: Structured Education Program

INTERVENTIONS:
Behavioral: Lifestyle & Behavioral Change Program — Participants in the weight loss arm will receive an intensive group-based behavioral weight loss program. In the first six months of the intervention, all participants in the weight loss arm will be given skill-based diet and exercise prescriptions for weight loss and will be taught specific cognitive and behavioral skills to assist in the modification of their eating and exercise habits. Participants will meet weekly for 6 months in group sessions led by a nutritionist, exercise physiologist, or behaviorist and will follow a structured protocol. This intervention strategy is modeled on interventions that have been successful in other overweight populations and is similar to the programs implemented in our ongoing studies, such as Look AHEAD. With this intervention, women are expected to lose on average of 7-9% of their initial body weight.
  Arms: Lifestyle & Behavioral Change Program
Behavioral: Structured Education Program — Women randomized to the Structured Education Program will be invited to participate in hour long group educational sessions at months 1, 2, 3, and 4. At months 6, 9 and 15, the groups will meet again for group support sessions. The content of these education and support sessions will include information about weight loss, physical activity, healthy eating habits and general health promotion. The educational sessions will be delivered primarily in a group format, with individual make up sessions provided for participants who miss group sessions.
  Arms: Structured Education Program

SUMMARY:
PRIDE will evaluate the impact of weight loss on urinary incontinence in a randomized, controlled trial.

DETAILED DESCRIPTION:
Three hundred and thirty overweight and obese women with urinary incontinence, 165 from each of two Clinical Centers, will be randomized to either a 6-month intensive behavioral weight control program or to usual care (no weight reduction intervention) and followed for 18 months. Efficacy of weight reduction as a treatment for urinary incontinence will be examined at 6 months following the intensive weight control program, and the sustained impact of the intervention will be examined at 18 months. To increase the maintenance of weight reduction and facilitate evaluation of the enduring impact of weight loss on urinary incontinence, we propose to study a motivation-based weight maintenance program. At the end of the intensive weight control program, women randomized to the weight loss program will be randomized to either a 12-month skill-based maintenance intervention or to a motivation-based maintenance intervention. The maintenance interventions maximize the potential for sustained weight loss and will allow us to determine if long-term weight reduction will produce continued improvement in urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 30 years and not institutionalized
* body mass index 25 to 50 kg/m2
* urinary incontinence symptoms for > 3 months by self-report and record > 10 incontinent episodes per week on a 7-day urinary diary
* able to complete a behavioral run-in consisting of self-monitoring of food and activity
* report having a primary health care provider
* able to understand and sign informed consent and complete baseline questionnaires
* agree to not initiate new treatment for incontinence or weight reduction, including behavioral, pharmacological or surgical therapies, for the duration of the study

Exclusion Criteria:

* current use, or use within the previous month of medical therapy for incontinence
* currently pregnant or gave birth in the previous 6 months
* current urinary tract infection (dipstick urinalysis positive for leukocyte esterase, nitrites or blood) or report having > 4 urinary tract infections in the preceding year
* incontinence of neurologic or functional origin (by history)
* self-report of prior anti-incontinence or urethral surgery, pelvic cancer or pelvic irradiation
* self-report of significant medical conditions of the genitourinary tract (genitourinary fistula, interstitial cystitis, symptomatic pelvic organ prolapse)
* report a medical condition that would affect the safety and/or efficacy of a weight management program involving diet and physical activity, including type 2 diabetes requiring medical therapy that may cause hypoglycemia, chronic steroid use or uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure > 100 mm Hg); women with a history of coronary heart disease may participate with written approval from their primary care physician
* currently engaged in an active weight loss program and/or experienced a 10% or greater weight reduction in the past 3 months
* report being unable to walk 2 blocks (1/4 mile) without stopping
* report conditions that, in the judgment of the Clinical Center Principal Investigator, render potential participants unlikely to follow the protocol for 18 months, including illness likely to be terminal within 2 years, plans to move, substance abuse or other significant psychiatric problems, or dementia
* participating in another research study that involves investigational drugs or can potentially confound the results of PRIDE

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in the number of incontinent episodes | 6 months
  Change in the number of incontinence episodes reported in a 7-day voiding diary from baseline to 6 months

SECONDARY OUTCOMES:
Change in body weight at 6 months | 6 months
  Change from baseline in body weight measured in kg
Change in body weight at 12 months | 12 months
  Change from baseline in body weight measured in kg
Change in body weight at 18 months | 18 months
  Change from baseline in body weight measured in kg

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, MD, PhD, Principal Investigator — UCSF Coordinating Center; Leslee Subak, MD, Principal Investigator — UCSF Coordinating Center; John Kusek, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Lee Nyberg, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - University of California at San Francisco, San Francisco, California
  - Miriam Hospital/Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/pride/?query=pride
URL: https://repository.niddk.nih.gov/studies/pride/?query=pride

REFERENCES:
- [Derived] Myers DL, Sung VW, Richter HE, Creasman J, Subak LL. Prolapse symptoms in overweight and obese women before and after weight loss. Female Pelvic Med Reconstr Surg. 2012 Jan-Feb;18(1):55-9. doi: 10.1097/SPV.0b013e31824171f9. PMID 22453270
- [Derived] Pinto AM, Subak LL, Nakagawa S, Vittinghoff E, Wing RR, Kusek JW, Herman WH, West DS, Kuppermann M. The effect of weight loss on changes in health-related quality of life among overweight and obese women with urinary incontinence. Qual Life Res. 2012 Dec;21(10):1685-94. doi: 10.1007/s11136-011-0086-2. Epub 2011 Dec 10. PMID 22161726
- [Derived] Pinto AM, Kuppermann M, Nakagawa S, Vittinghoff E, Wing RR, Kusek JW, Herman WH, Subak LL. Comparison and correlates of three preference-based health-related quality-of-life measures among overweight and obese women with urinary incontinence. Qual Life Res. 2011 Dec;20(10):1655-62. doi: 10.1007/s11136-011-9896-5. Epub 2011 Apr 3. PMID 21461953
- [Derived] West DS, Gorin AA, Subak LL, Foster G, Bragg C, Hecht J, Schembri M, Wing RR; Program to Reduce Incontinence by Diet and Exercise (PRIDE) Research Group. A motivation-focused weight loss maintenance program is an effective alternative to a skill-based approach. Int J Obes (Lond). 2011 Feb;35(2):259-69. doi: 10.1038/ijo.2010.138. Epub 2010 Aug 3. PMID 20680012
- [Derived] Wing RR, Creasman JM, West DS, Richter HE, Myers D, Burgio KL, Franklin F, Gorin AA, Vittinghoff E, Macer J, Kusek JW, Subak LL; Program to Reduce Incontinence by Diet and Exercise (PRIDE). Improving urinary incontinence in overweight and obese women through modest weight loss. Obstet Gynecol. 2010 Aug;116(2 Pt 1):284-292. doi: 10.1097/AOG.0b013e3181e8fb60. PMID 20664387
- [Derived] Wing RR, West DS, Grady D, Creasman JM, Richter HE, Myers D, Burgio KL, Franklin F, Gorin AA, Vittinghoff E, Macer J, Kusek JW, Subak LL; Program to Reduce Incontinence by Diet and Exercise Group. Effect of weight loss on urinary incontinence in overweight and obese women: results at 12 and 18 months. J Urol. 2010 Sep;184(3):1005-10. doi: 10.1016/j.juro.2010.05.031. PMID 20643425
- [Derived] Huang AJ, Subak LL, Wing R, West DS, Hernandez AL, Macer J, Grady D; Program to Reduce Incontinence by Diet and Exercise Investigators. An intensive behavioral weight loss intervention and hot flushes in women. Arch Intern Med. 2010 Jul 12;170(13):1161-7. doi: 10.1001/archinternmed.2010.162. PMID 20625026
- [Derived] Subak LL, Wing R, West DS, Franklin F, Vittinghoff E, Creasman JM, Richter HE, Myers D, Burgio KL, Gorin AA, Macer J, Kusek JW, Grady D; PRIDE Investigators. Weight loss to treat urinary incontinence in overweight and obese women. N Engl J Med. 2009 Jan 29;360(5):481-90. doi: 10.1056/NEJMoa0806375. PMID 19179316